CLINICAL TRIAL: NCT05700539
Title: A Randomized Controlled Trial of Internet-based Cognitive Behavioral Therapy for Adult Attention Deficit Hyperactivity Disorder in Sweden
Brief Title: Internet-based Cognitive Behavioral Therapy for Adult Attention Deficit Hyperactivity Disorder
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Karolinska Institutet (Other)
Collaborators: Uppsala University (Other)
Responsible Party: Principal Investigator, Alexander Rozental, Principal Investigator, Karolinska Institutet
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: DF0001
Record Dates: First submitted 2022-12-21; First posted 2023-01-26 (Actual); Last update posted 2025-09-02 (Actual); Status verified 2025-08

CONDITIONS: ADHD
MeSH Terms: conditions — Attention Deficit Disorder with Hyperactivity

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Internet-based cognitive behavioral therapy (Experimental)
  Interventions: Behavioral: Internet-based cognitive behavioral therapy
- Wait-list control (No Intervention)

INTERVENTIONS:
Behavioral: Internet-based cognitive behavioral therapy — A ten-week treatment based on cognitive behavioral therapy for ADHD, including two mandatory modules and at least four self-selected modules (out of ten available modules). The treatment consists of reading material and exercises to be completed each week.
  Arms: Internet-based cognitive behavioral therapy

SUMMARY:
Attention deficit hyperactivity disorder (ADHD) is a disorder characterized by lack of attention, hyperactivity, and impulsivity. It can have major impact on everyday life and result in negative consequences for one's personal, academic, and work situation. For individuals with symptoms of ADHD, increased levels of anxiety and depression are common, and an overall reduction of quality of life is often present. This study protocol describes a clinical trial of internet-based cognitive behavioral therapy (iCBT), using a randomized controlled study design, with the primary aim to increase quality of life, as well as to reduce symptoms of ADHD, anxiety, depression, and stress. A second aim is to investigate, by qualitative means, what aspects of treatment were perceived as helpful and hindering when it comes to completing iCBT. Two hundred participants with symptoms of ADHD will be included and randomized to two conditions (treatment and wait-list control). The treatment period is comprised of ten weeks, with two mandatory modules and ten modules from which the participants can choose freely. Self-report measures are completed by the participants at baseline and end of treatment, as well as at a six-month follow-up. The treatment is guided by therapists and consists of weekly correspondence with the participants. The study will utilize an intention to treat design, with ANOVAs and Reliable Change Index to evaluate treatment effects. The qualitative part of the project will be interview-based and employ thematic analysis. Lastly, a psychometric evaluation of a common instrument for determining ADHD-symptoms will also be made. The results will hopefully contribute to the evidence base for iCBT for individuals with symptoms of ADHD and help disseminate potentially effective interventions.

ELIGIBILITY:
Inclusion Criteria:

1. Over 18 years old of age.
2. Can read and write in Swedish.
3. Have access to a computer, tablet, or smartphone with an Internet connection.
4. Have previously been diagnosed with ADHD.
5. Are studying at a university or college in Sweden or working at least 50% of a full time-employment.

Exclusion Criteria:

1. Shows elevated symptoms of depression or risk of suicide, i.e., a total score on the Patient Health Questionnaire - 9 items (PHQ-9; Kroenke, K., Spitzer, R. L., & Williams, J. B. (2001)), > 15 points, or scores > 2 points on question i) concerning suicidality.
2. Has started or changed their medication for any psychiatric diagnosis in the last three months.
3. Exhibits another form of psychiatric diagnosis that requires more specialized care, for example substance abuse syndrome, anorexia nervosa, bipolar disorder, psychotic symptoms, or schizophrenia, as assessed with the MINI (Sheehan et al., 1998).

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 200 (Estimated)
Dates: Start 2023-01-25 (Actual); Primary Completion 2025-11-01 (Estimated); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
Adult Attention-deficit/hyperactivity disorder Quality-of-Life scale (AAQoL) | Change in quality of life from baseline to 10 week (i.e., post-treatment)
  The AAQoL (Brod et al., 2015; Brod, Johnston, Able, & Swindle, 2006) is a disease-specific quality of life measure for adults with ADHD. The instrument measures quality of life-consequences of ADHD in four domains using and consists of 29 items. The instrument has excellent internal consistency (Cronbach's α = .93 for the overall measure). One example of an item is "In the last two weeks, how hard has it been for you to remember important things?", scored on a five-point Likert-like scale from "Not at all/Never" (1) to "Extremely/Very Often" (5). The scale ranges from 0 to 145.
Adult Attention-deficit/hyperactivity disorder Quality-of-Life scale (AAQoL) | Change in quality of life from baseline six-month follow-up
  The AAQoL (Brod et al., 2015; Brod, Johnston, Able, & Swindle, 2006) is a disease-specific quality of life measure for adults with ADHD. The instrument measures quality of life-consequences of ADHD in four domains using and consists of 29 items. The instrument has excellent internal consistency (Cronbach's α = .93 for the overall measure). One example of an item is "In the last two weeks, how hard has it been for you to remember important things?", scored on a five-point Likert-like scale from "Not at all/Never" (1) to "Extremely/Very Often" (5). The scale ranges from 0 to 145.
Adult ADHD Self-Report Scale-V1.1 (ASRS-V1.1) Symptoms Checklist (ASRS) | Change in ADHD symptoms from baseline to 10 week (i.e., post-treatment)
  The ASRS is an instrument that measures ADHD-symptoms (Kessler et al., 2005). The instrument consists of 18 items that correspond to the 18 symptom-criteria for ADHD found in the DSM-IV-TR (Association, 2000). Of these 18 questions, six have been identified as most predictive of ADHD-symptoms. The overall range of the entire measure is 0 to 72. However, there are separate items focusing on attention and hyperactivity.
Adult ADHD Self-Report Scale-V1.1 (ASRS-V1.1) Symptoms Checklist (ASRS) | Change in ADHD symptoms from baseline to six-month follow-up
  The ASRS is an instrument that measures ADHD-symptoms (Kessler et al., 2005). The instrument consists of 18 items that correspond to the 18 symptom-criteria for ADHD found in the DSM-IV-TR (Association, 2000). Of these 18 questions, six have been identified as most predictive of ADHD-symptoms. The overall range of the entire measure is 0 to 72. However, there are separate items focusing on attention and hyperactivity.

SECONDARY OUTCOMES:
Generalized Anxiety Disorder - 7 Items (GAD-7) | Change in anxiety symptoms from baseline to 10 week (i.e., post-treatment)
  The GAD-7 is an instrument that measures anxiety (Spitzer, Kroenke, Williams, & Löwe, 2006). Its internal consistency is excellent (Cronbach's α = .92), and it has good test-retest reliability (IntraClass Correlation = .83; Spitzer et al., 2006). The instrument includes seven items and has a single-factor solution. The score ranges from 0 to 21 points and the items range from 0 ("Not at all") to 3 ("Nearly every day"; Spitzer et al., 2006). One example of an item is: "Over the last 2 weeks, how often have you been bothered by any of the following problems? Feeling nervous, anxious, or on edge."
Generalized Anxiety Disorder - 7 Items (GAD-7) | Change in anxiety symptoms from baseline to six-month follow-up
  The GAD-7 is an instrument that measures anxiety (Spitzer, Kroenke, Williams, & Löwe, 2006). Its internal consistency is excellent (Cronbach's α = .92), and it has good test-retest reliability (IntraClass Correlation = .83; Spitzer et al., 2006). The instrument includes seven items and has a single-factor solution. The score ranges from 0 to 21 points and the items range from 0 ("Not at all") to 3 ("Nearly every day"; Spitzer et al., 2006). One example of an item is: "Over the last 2 weeks, how often have you been bothered by any of the following problems? Feeling nervous, anxious, or on edge."
Patient Health Questionnaire - 9 Items (PHQ-9) | Change in depressive symptoms from baseline to 10 week (i.e., post-treatment)
  The PHQ-9 is a nine-item instrument measuring depression. It has excellent internal consistency (Cronbach's α = .89) and a good test-retest correlation (r = .84; Kroenke et al., 2001). The instrument has a single-factor solution. The score ranges from 0 to 27 points (Kroenke, Spitzer, & Williams, 2001). Items range from 0 ("Not at all") to 3 ("Nearly every day"). One example of an item is: "Over the last 2 weeks, how often have you been bothered by any of the following problems? Little interest or pleasure in doing things."
Patient Health Questionnaire - 9 Items (PHQ-9) | Change in depressive symptoms from baseline to six-month follow-up
  The PHQ-9 is a nine-item instrument measuring depression. It has excellent internal consistency (Cronbach's α = .89) and a good test-retest correlation (r = .84; Kroenke et al., 2001). The instrument has a single-factor solution. The score ranges from 0 to 27 points (Kroenke, Spitzer, & Williams, 2001). Items range from 0 ("Not at all") to 3 ("Nearly every day"). One example of an item is: "Over the last 2 weeks, how often have you been bothered by any of the following problems? Little interest or pleasure in doing things."
Perceived Stress scale (PSS) | Change in stress symptoms from baseline to 10 week (i.e., post-treatment)
  The PSS is an instrument that evaluates the subjective experience of general stress in various situations and is scored on a five-point Likert-scale 0-4 ("Never" to "Very often"), with seven items being scored in reverse (items 4-7, 9-10, and 13). The PSS includes 14 items in total and has been shown to have good internal consistency (Cronbach's α = .84-.86) as well as good convergent and discriminant validity (Cohen, Kamarck, & Mermelstein, 1983).
Perceived Stress scale (PSS) | Change in stress symptoms from baseline to six-month follow-up
  The PSS is an instrument that evaluates the subjective experience of general stress in various situations and is scored on a five-point Likert-scale 0-4 ("Never" to "Very often"), with seven items being scored in reverse (items 4-7, 9-10, and 13). The PSS includes 14 items in total and has been shown to have good internal consistency (Cronbach's α = .84-.86) as well as good convergent and discriminant validity (Cohen, Kamarck, & Mermelstein, 1983).
Negative Effects Questionnaire (NEQ) | Incidence of negative effects of psychological treatment from baseline to post-treatment
  The NEQ is a 32-item instrument that assesses unwanted and adverse events experienced by patients undergoing psychotherapy (Rozental, Kottorp, Boettcher, Andersson, & Carlbring, 2016; Rozental et al., 2019), e.g., "I experienced more unpleasant feelings". It is comprised of six factors: symptoms, quality, dependency, stigma, hopelessness, and failure. The internal consistency for the full instrument is excellent (Cronbach's α = .95), and is scored on several dimensions; 1) "Did you experience this?" (yes/no), 2) "If yes - here is how negatively it affected me", from 0 ("Not at all") to 4 ("Extremely"), and 3) "Probably caused by" ("The treatment I received" or "Other circumstances").

CONTACTS AND LOCATIONS:
Overall Officials: David Forsström, PhD, Principal Investigator — Uppsala University
Locations (1):
- Uppsala University, Uppsala, Sweden

IPD SHARING:
Plan to Share IPD: No